CLINICAL TRIAL: NCT02457234
Title: Examining the Influence of Cultural Immersion on Willingness to Try Fruits and Vegetables Among Children in Guam: the Traditions Study
Brief Title: Influence of Cultural Immersion on Willingness to Try Fruits and Vegetables Among Children in Guam: the Traditions Study
Acronym: Traditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guam (Other)
Collaborators: University of Hawaii (Other)
Responsible Party: Principal Investigator, Tanisha Aflague, Doctoral Candidate - CHL program, University of Guam
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CHRS #14-55
Record Dates: First submitted 2015-05-27; First posted 2015-05-29 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Food Preferences
Keywords: fruits and vegetables; cultural immersion
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cultural Immersion Children's Day Camp (Experimental): Participants in this group received four culturally adapted nutrition lessons within a cultural immersion context as part of the camp program.
  Interventions: Behavioral: Cultural immersion
- University Children's Day Camp (Active Comparator): Participants in this group received four culturally adapted nutrition lessons in addition to camp activities that did not include cultural immersion.
  Interventions: Behavioral: Cultural immersion
- Recreational Children's Sports Day Camp (No Intervention): Participants in this group participated in existing camp activities that were exclusively physical activity.

INTERVENTIONS:
Behavioral: Cultural immersion — The primary intervention was the cultural immersion within CIC. Unique to the Traditions study were culturally-adapted nutrition lessons incorporated into CIC and UDC. CIC had a high cultural dose as the Traditions lessons were implemented within the cultural immersion context of the camp. The UDC had moderate cultural dose from the Traditions lessons only. RSC was without cultural immersion and Traditions lessons or had zero cultural dose.
  Other Names: Culturally adapted nutrition lessons
  Arms: Cultural Immersion Children's Day Camp; University Children's Day Camp

SUMMARY:
The purpose of the Traditions study was to examine the influence of cultural immersion on willingness to try fruits and vegetables among children, 3-12 y, in Guam. The primary objective of this study was to examine willingness to try fruits and vegetables and fruit and vegetable intake among children attending three existing summer camp programs: a cultural immersion camp, a university day camp, and a recreational sports camp. The primary hypothesis was that children attending the cultural immersion camp would have higher willingness to try fruits and vegetables (WillTry score) and a higher intake of fruits and vegetables compared to children attending both, the university day camp and recreational sports camp, without cultural immersion.

A pre-post, quasi-experimental design was used to evaluate 3 summer camps with different exposure levels of cultural immersion. High, moderate, and zero (cultural) exposure was provided by a cultural immersion camp (CIC), a university-based day camp (UDC), and a recreational sports camp (RSC), respectively. CIC delivered 4 culturally adapted nutrition lessons within the context of Chamorro cultural traditions as part of the cultural immersion camp activities. The UDC delivered the same lessons within a physiology framework. The RSC was without nutrition lessons and cultural immersion. Children 3-12 years old registered in any of the three summer camp programs were eligible to participate. Data collection was primarily administered at two assessment periods: before (± 2 weeks) and after (± 1 week) each summer camp program. Children's willingness to try fruits and vegetables, the primary outcome, was assessed with the interview-administered Adapted WillTry tool. The secondary outcome was fruit and vegetable intake as servings/day in the CIC to UDC only. Fruit and vegetable intake was assessed using the mobile food record (mFR), which is an app running on an iPod Touch based on the technology assisted dietary assessment (TADA) protocols. Outcomes examined Adapted WillTry post-scores for local novel and local common fruits and vegetables and fruit and vegetable servings/day using multivariate regression models adjusting for the relevant pre-score, sex, age, ethnicity, dose, BMI percentile, and parent's cultural affiliation. Therefore, additional measures like sociodemographic information, anthropometry (i.e. heights and weights), and parent's cultural affiliation were collected to account for potential confounders.

DETAILED DESCRIPTION:
A pre-post quasi-experimental design was used to observe outcomes (i.e., willingness to try FV and FV intake) between three existing summer camp programs in Guam: cultural immersion camp (CIC), university day camp (UDC), and recreational sports camp (RSC). This natural-setting, multi-arm parallel design was used as an alternative to a resource intensive infrastructure and the organizations were willing to incorporate activities to answer the research question.

The CIC and UDC programs were nearly matched for daily activities (e.g., physical activity, cooking demonstrations/taste testing, crafts). The same four Traditions lessons (Figure 1) were incorporated into CIC and UDC and delivered by the same educators. These lessons featured local FV and promoted positive associations with eating FV. In CIC, the context of Chamorro cultural traditions, practices, and values was tied to FV. Chamorro is the language, culture, and ethnicity of Guam and the Marianas. In UDC, consuming healthy foods was introduced within a context of nutrition and human physiology. The four lessons were adapted with permission from a culturally-relevant Hawai'ian nutrition curriculum to make them relevant to Guam and the Chamorro culture. This curriculum complemented Hawai'i and Guam Department of Education K-12 Content and Performance Standards.

The CIC activities perpetuated the Chamorro culture and language through song/chanting, dance, prayer, arts and crafts, cooking, outdoor activities, and gardening based on traditional and contemporary practices. Chamorro was spoken about 80% of the time, including the delivery of key messages in the Traditions lessons. All activities operated on indigenous values of respect, love, humility, reciprocity, and camaraderie. The UDC activities focused on promoting healthful present-day recreational activities and global foods. The activities were an extension of the Expanded Food and Nutrition Education Program mission. RSC was exclusively physical activity. Upon completion of the last assessments, educators provided one Traditions lesson for registrants at RSC.

Data collection occurred at two assessment periods: before (± 2 weeks) and after (± 1 week) each program. The first assessment was completed at each camp setting. The second was also completed at camp or at a pre-arranged location, such as the children's home or a child-friendly public space (e.g., the mall). Children completed the interview-administered Adapted WillTry tool, which measures children's willingness to try FV and was previously validated for children 3-11 years old in Guam. FV intake was assessed using the mobile food record (mFR). The mFR is an app that has been shown to be a useful method for dietary assessment with adolescents. Only participants in CIC and UDC were asked to use the mFR due to a limited number of iPods.

Other Measures: Parents completed a questionnaire that included information about the child's age, sex, language spoken, religion, and birthplace. Parent's cultural affiliation was determined using their responses reported on a cultural affiliation questionnaire, which assesses one of four modes of acculturation: traditional, integrated, assimilated, or marginalized. The same scoring system was used as described by Kaholokula and others. Anthropometric assessments were completed at a time designated as least disruptive to camp activities. Height and weight were measured using a portable Seca scale and stadiometer (PE-AIM 101) using centimeters and kilograms, respectively. These measurements were converted to body mass index (BMI) as [kg/(height, m)2]. Dose was assessed by recording attendance at camp and at each Traditions lesson.

For participation, all children were given a gift card, in $5 or $10 denominations, one before and one after camp assessments. Remuneration varied due to the different types and lengths of involvement for participants depending on camp program.

Sample size was determined using estimates for the Adapted WillTry local novel and local common FV scores from data representing children similar to children recruited for this study. The main outcomes, model 1 and model 2 were powered at 0.8 for a minimum detectable difference (MDD) of 0.43 for the local novel score and 0.41 for the local common score which corresponded to proposed sample sizes of n=60 for CIC, n=30 for UDC, and n=30 for RSC. For Model 3, based on the UDC and RSC sample sizes MDD was 0.49 and 0.47 for local novel and local common, respectively. For the secondary outcome, post-FV intake, the MDDs were 0.877, 0.3132, and 0.6265 per day dependent on the baseline FV consumption being 2, 1 or 1.5 which yielded sample sizes for CIC (n=60) and UDC (n=30).

Data were entered using a Microsoft Access (Microsoft Corp) tool specifically designed for this study. Double-data entry procedures were used and PROC COMPARE in SAS 9.3 (SAS Institute, Inc.) was performed until both data entries achieved 100% matching. A trained analyst examined images, identified all whole FV (e.g., FV mixed dishes, fruits, vegetables), and amounts consumed. FV (100%) juices were excluded. FV intake was calculated by dividing the total FV by the total number of days eating occasions were captured using the mFR.

Categorical variables were examined using frequencies and for quantitative variables means and standard deviations were used. Differences between camps in Adapted WillTry FV post-scores (i.e. local novel, local common, and imported) were examined using univariate ANOVA adjusted for pre-scores. To examine the previously observed incremental trend of the Adapted WillTry FV scores, where each score was statistically significantly different from one another, the paired t-tests for each pre- and post-assessment score in all camps were performed. Analytical analyses were conducted using IBM SPSS Statistics version 21 (IBM Corporation, Armonk, NY).

Potential confounders were included in models using indicator variables for age (i.e., 3-6y, 7-8y, 9-12y), ethnicity (i.e., Chamorro, Chamorro Mixed, Other), and sex. Categories of parent's cultural affiliation were analyzed as traditional and integrated. In these models, children whose parents were categorized as marginalized (n=2) or assimilated (n=1) were eliminated due to small numbers. Lesson and camp attendance dose for CIC and UDC were calculated using the sum of days participants attended lessons and camp days divided by the total possible lesson and camp days, respectively. A dichotomous variable was created for high and low dose using the 50th percentile cut-point for lessons and camp dose. BMI was modeled as a continuous variable.

To examine the primary hypothesis, indicator variables were created for each camp for relevant comparisons in Models 1, 2, and 3. Multiple linear regression models for the three Adapted WillTry post-scores (dependent variables) were fit separately to examine whether and how much the Adapted WillTry scores differed by camp program accounting for potential confounders (i.e., pre-scores, participant's age, sex, ethnicity, BMI, parent's cultural affiliation, and lesson and camp days dose). The final model included Adapted WillTry pre-scores, sex, age, and ethnicity. For whole FV intake, multiple linear regression models were used to examine differences in post-FV intake/day (dependent variable) between UDC and CIC. The final model included pre-FV intake/day, age, ethnicity, and parent's cultural affiliation (independent variables).

ELIGIBILITY:
Inclusion Criteria:

* Summer camps over 4 weeks serving children 3-12 years old in Guam

Exclusion Criteria:

* Summer camps shorter or greater than 4 weeks serving children older than 12 years old in Guam

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Willingness to try local fruits and vegetables measured by the Adapted WillTry tool. | 4 weeks
  The Adapted WillTry tool measures children's willingness to try FV and was previously validated for children 3-11 years old in Guam. The Adapted WillTry has 3 distinct scales of FV: local novel, local common, and imported. The scores for each scale ranged from 1 to 3, i.e., least to most willing to try. The Adapted WillTry administration and scoring methods have been described previously.

SECONDARY OUTCOMES:
Fruit and vegetable intake measured using the mobile food record | 4 weeks
  FV intake was assessed using the mobile food record (mFR) running on iOS7.1.2 on an Apple iPod touch. Only participants in CIC and UDC were asked to use the mFR due to a limited number of iPods. Children used the mFR for two consecutive days to capture before and after images of all eating occasions. Instructions on how to use the mFR included taking a practice image of plastic food replicas with a fiducial marker (FM). The FM functioned as a color reference and volume marker of the food. Children were loaned the mFR and 2-4 FMs. When the children returned the mFR, researchers asked children to assist with identifying food items that were indistinguishable, e.g., opaque containers, occluded foods; and to recall foods at eating occasions not captured as an image.

CONTACTS AND LOCATIONS:
Overall Officials: Carol J Boushey, PhD, Study Chair — University of Hawaii Cancer Research Center

REFERENCES:
- [Background] Blanchette L, Brug J. Determinants of fruit and vegetable consumption among 6-12-year-old children and effective interventions to increase consumption. J Hum Nutr Diet. 2005 Dec;18(6):431-43. doi: 10.1111/j.1365-277X.2005.00648.x. PMID 16351702
- [Background] Aflague TF, Leon Guerrero RT, Boushey CJ. Adaptation and evaluation of the WillTry tool among children in Guam. Prev Chronic Dis. 2014 Aug 21;11:E142. doi: 10.5888/PCD11.140032. PMID 25144677
- [Background] Thomson JL, McCabe-Sellers BJ, Strickland E, Lovera D, Nuss HJ, Yadrick K, Duke S, Bogle ML. Development and evaluation of WillTry. An instrument for measuring children's willingness to try fruits and vegetables. Appetite. 2010 Jun;54(3):465-72. doi: 10.1016/j.appet.2010.01.012. Epub 2010 Jan 29. PMID 20116407
- [Background] Six BL, Schap TE, Zhu FM, Mariappan A, Bosch M, Delp EJ, Ebert DS, Kerr DA, Boushey CJ. Evidence-based development of a mobile telephone food record. J Am Diet Assoc. 2010 Jan;110(1):74-9. doi: 10.1016/j.jada.2009.10.010. PMID 20102830
- [Background] Daugherty BL, Schap TE, Ettienne-Gittens R, Zhu FM, Bosch M, Delp EJ, Ebert DS, Kerr DA, Boushey CJ. Novel technologies for assessing dietary intake: evaluating the usability of a mobile telephone food record among adults and adolescents. J Med Internet Res. 2012 Apr 13;14(2):e58. doi: 10.2196/jmir.1967. PMID 22504018
- [Background] Renzaho AM, Swinburn B, Burns C. Maintenance of traditional cultural orientation is associated with lower rates of obesity and sedentary behaviours among African migrant children to Australia. Int J Obes (Lond). 2008 Apr;32(4):594-600. doi: 10.1038/ijo.2008.2. Epub 2008 Feb 5. PMID 18253161
- [Background] Kuhnlein H, Erasmus B, Creed-Kanashiro H, Englberger L, Okeke C, Turner N, Allen L, Bhattacharjee L. Indigenous peoples' food systems for health: finding interventions that work. Public Health Nutr. 2006 Dec;9(8):1013-9. PMID 17125565